CLINICAL TRIAL: NCT03975296
Title: Transmuscular Quadratus Lumborum Block Versus Thoracic Paravertebral Block for Acute Pain and Quality of Recovery After Laparoscopic Partial Nephrectomy
Brief Title: QLB Versus PVB for Acute Pain and Quality of Recovery After Laparoscopic Partial Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cui Xulei (Other)
Responsible Party: Sponsor-Investigator, Cui Xulei, The attending physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CXL3
Record Dates: First submitted 2019-06-02; First posted 2019-06-05 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2020-03

CONDITIONS: Nerve Block, Nephrectomy, Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMQLB group (Experimental)
  Interventions: Procedure: preoperative single-shot TMQLB; Drug: patient controlled intravenous analgesia(PCIA)
- TPVB group (Active Comparator)
  Interventions: Procedure: preoperative single-shot TPVB; Drug: patient controlled intravenous analgesia(PCIA)

INTERVENTIONS:
Procedure: preoperative single-shot TMQLB — The patient is placed in the lateral position. The curved probe of Ultrasound Scanner is used for scan and located vertical to the iliac crest at the posterior axillary line to find the Shamrock sign. The 22-G needle is then inserted in plane and directed to the QL muscle. After the proper position of the needle tip between the psoas major muscle and the quadratus lumborum muscle is confirmed, 0. 6 ml/kg 0.5% ropivacaine is injected into the interfascial plane.
  Followed by IPCA in the first 48h after surgery: morphine boluses: 1.5-2 mg, lockout time :10 min, 1h limitation: 6-8 mg morphine.
  Arms: TMQLB group
Procedure: preoperative single-shot TPVB — The patient is placed in the lateral position, the spinous processes of T10 are identified and marks are made 2cm lateral to the spinous processes. The curve probe of ultrasound scanner is placed transversally at the mark to identify the paravertebral space. Then a 22-G needle is inserted in-plane from lateral to medial and advanced until the tip reached the paravertebral space surrounded by the parietal pleura and the superior costotransverse ligament. 0.4 ml/kg 0.5% ropivacaine is injected into the paravertebral space of T10.
  Arms: TPVB group
Drug: patient controlled intravenous analgesia(PCIA) — at the end of surgery, patient is administered a PCIA with morphine boluses: 1.5-2 mg, lockout time :10 min, 1h limitation: 6-8 mg morphine.

SUMMARY:
This trial is a prospective, randomized, single-center, open-label, parallel-arm, blinded-analysis trial, the objective of which is to evaluate the effect of transmuscular quadratus lumborum block (TMQLB) in the pain relief and quality of recovery in laparoscopic partial nephrectomy compared with thoracic paravertebral block (TPVB).

ELIGIBILITY:
Inclusion Criteria:

Age 18-70 yrs American Society of Anesthesiologists physical statusⅠ-Ⅲ Undergo laparoscopic nephrectomy Informed consent

Exclusion Criteria:

A known allergy to the drugs being used Coagulopathy, on anticoagulants Analgesics intake, history of substance abuse Participating in the investigation of another experimental agent Inability to properly describe postoperative pain to investigators (eg, language barrier, neuropsychiatric disorder)

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
cumulative morphine consumption | within 48 postoperative hours

SECONDARY OUTCOMES:
The pain scores determined by the numeric rating scale (NRS, 0-10) | within 48 postoperative hours
  NRS is an internationally recognized pain scale with 11 points ranging from 0 to 10 points, with 0 defined as no pain and 10 defined as the worst pain imaginable.
dermatomal distribution of sensory reduction | 30 min after the block
  Thirty minutes after the block, the bilateral dermatomal sensory blocks for the anterior abdomen (between the anterior axillary and mid-clavicular lines) and thigh were assessed with the pinprick method. A reduce in pinprick sensation relative to the unblocked side was interpreted as an effective block.
quality of recovery evaluated by the self-assessment 15-item quality of recovery (QoR) scale | at 3 days and 5 days after the sugery
  QoR is a 15-item questionnaire which will score on a scale of 0-10 pertaining to patient's comfort, support system, pain, well-being, and ability to carry out daily activities, where 0 indicates none of the time and 10 indicates all of the time
postoperative length of hospital stay | within 2 weeks after the surgery
  time to patient's discharge
patient satisfaction with anesthesia | 48 hours after surgery
  use the Chinese version Bauer questionnaire to assess the patient satisfaction with anesthesia
nausea and vomiting episodes | within 24 hours after the surgery]
ambulation time | within the 5 days after surgery
  time from the end of the surgery to the first time to out-of-bed activity
time of recovery of bowl movement | within the 5 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: yuguang huang, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Wang J, Cui X, Ren L, Li X, Zhang Y, Xie Y, Ji Z, Huang Y. Comparison of the Postoperative Analgesic Effects between Ultrasound-Guided Transmuscular Quadratus Lumborum Block and Thoracic Paravertebral Block in Laparoscopic Partial Nephrectomy Patients: A Randomized, Controlled, and Noninferiority Study. Pain Res Manag. 2023 Feb 20;2023:8652596. doi: 10.1155/2023/8652596. eCollection 2023. PMID 36891030